CLINICAL TRIAL: NCT04943874
Title: Feasibility and Acceptability of a Biofeedback Based Virtual Reality Intervention to Manage Postoperative Pain in Children and Adolescents After Surgery
Brief Title: Biofeedback Based Virtual Reality Intervention to Manage Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanessa Olbrecht (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Vanessa Olbrecht, Chair, Department of Anesthesiology & Perioperative Medicine, Nemours Children's Clinic
Organization: Nemours Children's Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-0994; 5R34AT011218 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-06-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pain; Pain, Postoperative; Pain, Acute; Surgery
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Technology Based Intervention 1 (Phase 1) (Other)
  Interventions: Device: Technology Based Intervention Group 1
- Technology Based Intervention 1 (Phase 2) (Other)
  Interventions: Device: Technology Based Intervention Group 1
- Technology Based Intervention 2 (Phase 2) (Other)
  Interventions: Device: Technology Based Intervention Group 2

INTERVENTIONS:
Device: Technology Based Intervention Group 1 — In Phase 1, all participants will use the same technology. In Phase 2, participants will be blinded to the two specific groups. They will not be aware of the technology used in the group they are not assigned too.
  Arms: Technology Based Intervention 1 (Phase 1); Technology Based Intervention 1 (Phase 2)
Device: Technology Based Intervention Group 2 — Participants will be blinded to the two specific groups. They will not be aware of the technology used in the group they are not assigned too.
  Arms: Technology Based Intervention 2 (Phase 2)

SUMMARY:
To develop and refine a technology based treatment protocol for preoperative education and training and postoperative care in children and adolescents undergoing surgery.

DETAILED DESCRIPTION:
This is a 2-phase study aimed to refine a perioperative treatment protocol for a technology-based intervention (Aim 1) and to understand whether technology-based interventions can be used to help treat pain in children following surgery (Aim 2). Patients will participate in only one phase of the study, and when patients are enrolled will determine what Phase of the study they are in.

In Phase 1, all patients will use the same technology, and no randomization will occur. Primary and secondary outcome measures of Aim 1 are assessed in Phase 1. Actual enrollment for Phase 1 was 23 patients.

In Phase 2, patients will be randomized to receive 1 of 2 technology-based interventions. The perioperative treatment protocol developed in Phase 1 (Aim 1) will be used in Phase 2 to assess the primary and secondary outcome measures of Aim 2. This phase is anticipated to enroll up to 70 participants.

This is not an FDA-regulated drug or device trial as the technology used in this study is categorized as a relaxation device by the FDA and considered "minimal risk", thus exempt from both NDE and IDE.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 -18 years
* Scheduled to undergo surgery anticipated to cause moderate to severe pain with expected length of stay > or = to 2 days
* Able to read, understand and speak English
* Patients requiring management by the Acute Pain Service
* Possession of a mobile device/computer available for study participation

Exclusion Criteria:

* Outside the age range (< 12 or > 18 years)
* Non-English speaking
* History of significant developmental delay, uncontrolled psychiatric conditions associated with hallucinations or delusions, or neurological conditions (especially epilepsy and/or significant motion sickness/nausea/vomiting)
* History of vertigo, dizziness, seizure disorder, and/or severe motion sickness
* History of chronic pain
* Are chronically using opioids and or benzodiazepines for the management of pain
* Are actively experiencing nausea or vomiting
* Conditions such as craniofacial abnormalities or surgeries of the head and neck
* Previous participation in this study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Aim 1: Treatment protocol refinement | Duration of study up to 30 days
  Frequency of sessions
Aim 1: Treatment protocol refinement | Duration of study up to 30 days
  Duration of sessions
Aim 2: Feasibility of technology intervention in perioperative patients | Pre-intervention
  Rate of study recruitment

SECONDARY OUTCOMES:
Aim 1: Preoperative training protocol | Up to two weeks pre-operatively
  Frequency of preoperative training session
Aim 1: Preoperative training protocol | Up to two weeks pre-operatively
  Duration of preoperative training session
Aim 1: Post-operative session protocol | Up to two week post surgery
  Frequency of post-operative intervention session
Aim 1: Post-operative session protocol | Up to two weeks post surgery
  Duration of post-operative intervention session
Aim 2: Rate of study enrollment/randomization | Pre-intervention
  Assessment of ability to enroll and randomize patients in pilot clinical trial
Aim 2: Rate of study retention | Duration of study up to 30 days
  Assessment of ability to retain patients in pilot clinical trial
Aim 2: Rate of treatment adherence | Duration of study up to 30 days
  Assessment of patient adherence to study protocol
Aim 2: Treatment-specific satisfaction | Post intervention up to two weeks
  Qualitative feedback from participants using questionnaire to assess intervention satisfaction
Aim 2: Treatment-specific satisfaction | Post intervention up to two weeks
  Qualitative feedback from participants using semi-structured interview to assess intervention satisfaction
Aim 2: Effect of technology on anxiety | 30 minutes after using technology
  Anxiety scores will be collected. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Aim 2: Effect of technology on medication use | Duration of hospital stay (2-7 days)
  Medications used will be collected
Aim 2: Effect of technology on anxiety | Before using technology
  Anxiety scores will be collected. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Aim 2: Effect of technology on anxiety | Immediately after using technology
  Anxiety scores will be collected. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Aim 2: Effect of technology on pain | Preoperatively (up to 5 days)
  Pains scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Aim 2: Effect of technology on pain | Before using technology
  Pains scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Aim 2: Effect of technology on pain | Immediately after using technology
  Pains scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Aim 2: Effect of technology on pain | 30 minutes after using technology
  Pains scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Aim 2: Self-Reported Outcomes | Day of hospital discharge (Postoperatively 2-7 days)
  Semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Olbrecht, MD, Principal Investigator — Nemours Children's Hospital
Locations (1):
- Nemours Children's Hospital, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with the public, but aggregate data will be publicly available upon request.

REFERENCES:
- [Derived] Orgil Z, Karthic A, Bell NF, Heisterberg LM, Williams SE, Ding L, Kashikar-Zuck S, King CD, Olbrecht VA. Use of Biofeedback-Based Virtual Reality in Pediatric Perioperative and Postoperative Settings: Observational Study. JMIR Perioper Med. 2024 Sep 16;7:e48959. doi: 10.2196/48959. PMID 38742940
- [Derived] Orgil Z, Johnson L, Karthic A, Williams SE, Ding L, Kashikar-Zuck S, King CD, Olbrecht VA. Feasibility and acceptability of perioperative application of biofeedback-based virtual reality versus active control for pain and anxiety in children and adolescents undergoing surgery: protocol for a pilot randomised controlled trial. BMJ Open. 2023 Jan 25;13(1):e071274. doi: 10.1136/bmjopen-2022-071274. PMID 36697053

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04943874/Prot_SAP_000.pdf